CLINICAL TRIAL: NCT04390048
Title: Balance Training With Transcranial Direct Current Stimulation (tDCS) for Chronic Ankle Instability (CAI)
Brief Title: Balance Training With tDCS for CAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Brian Arwari, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20200090
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Ankle Injuries and Disorders
Keywords: Chronic Ankle Instability
MeSH Terms: conditions — Ankle Injuries; Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Anodal tDCS and Balance Training (BT) Group (Experimental): Participants will undergo 4 weeks of BT under anodal tDCS treatment.
  Interventions: Device: Anodal tDCS
- Sham tDCS and BT Group (Sham Comparator): Participants will undergo 4 weeks of BT under sham tDCS.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Anodal tDCS — An anodal surface electrode will be attached to the contralateral motor cortex (M1) of the CAI-involved side and the reference electrode will be placed on the ipsilateral side of the supraorbital ridge. Anodal tDCS will deliver a low electrical current stimulation at 2 milliamps (mA). Participants will undergo 3 sessions per week for a total of 12 sessions and each session will last approximately 20 minutes.
  Arms: Anodal tDCS and Balance Training (BT) Group
Device: Sham tDCS — An anodal surface electrode will be attached to the contralateral motor cortex (M1) of the CAI-involved side and the reference electrode will be placed on the ipsilateral side of the supraorbital ridge. Sham tDCS will deliver a low electrical current stimulation at 2 mA and will be turned off 30 seconds following the application. Participants will undergo 3 sessions per week for a total of 12 sessions and each session will last approximately 20 minutes.
  Arms: Sham tDCS and BT Group

SUMMARY:
The purpose of this research study is to examine the efficacy of non-invasive brain stimulation in addition to balance exercise for chronic ankle instability (CAI), a condition that develops following an initial ankle sprain, usually because of loose or unstable ankle joints.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be neurologically sound
* Subjects should have abilities to maintain a single-leg stance at least for 10 seconds.
* A history of ankle sprain
* A history of ankle joint giving ways
* Current feelings of ankle joint instability

Exclusion Criteria:

* Individuals with a clinically defined neurological disorder, with an increased risk of seizure for any reason, with a history of treatment with Transcranial Magnetic Stimulation (TMS), deep brain stimulation for any disorder will be excluded.
* Patients with cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed will be excluded.
* A history of balance or vestibular disorder
* A history of previous surgeries to the musculoskeletal structures in either limb of the lower extremity
* A history of a fracture in either limb of the lower extremity requiring realignment
* A history of acute injuries to the lower extremity joints in the previous 3 months, which impacted joint integrity and function (i.e., sprains, fractures) resulting in at least 1 interrupted day of desired physical activity
* A history of herniated disc
* Poorly controlled headache
* Hypersensitivity to electrical or magnetic stimulation
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoner

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Arwari, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 24 participants signed informed consent and were enrolled in the study; however, 5 participants withdrew due to scheduling conflicts that occurred after participant enrollment, but prior to assignment of participants to an arm or group; therefore, the enrollment number in the protocol section will differ from the results section as 5 participants did not receive the intervention. The unit assignment are whole participants that have been assigned to the arms/groups.
Period: Overall Study
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Started | 10 | 9
Completed | 9 | 6
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.1 (8.2) | 22.3 (6.7) | 22.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 4 | 2 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 15
Height [Mean (Standard Deviation); unit: cm] | 173.6 (9.8) | 170.6 (9.7) | 172.4 (9.5)

OUTCOME MEASURES:

1. Primary Outcome: Static Postural Balance
Description: Center of Pressure (COP) velocity (cm/s)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: CM/S
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 9 | 6
CM/S | 57.0 (3.6) | 55.9 (3.7)

2. Primary Outcome: Static Postural Balance
Description: Center of Pressure (COP) velocity (cm/s)
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: CM/S
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 9 | 6
CM/S | 3.4 (0.7) | 3.4 (0.7)

3. Primary Outcome: Active Motor Threshold (AMT)
Description: The active motor threshold (AMT) was measured by transcranial magnetic stimulation (TMS) using a computation program, Parameter Estimation by Sequential Testing (PEST). AMT was defined as the minimum TMS intensity required to elicit an adequate motor-evoked potential (MEP) in the soleus muscle. A lower AMT reflects greater corticospinal excitability. The unit of measure is Percentage of Maximum Stimulus Output (MSO)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percentage of MSO
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 8 | 5
Percentage of MSO | 43.6 (9.0) | 39.4 (13.1)

4. Primary Outcome: Active Motor Threshold (AMT)
Description: as for outcome 3
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Percentage of MSO
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 8 | 5
Percentage of MSO | 43.9 (12.1) | 39.4 (13.0)

5. Secondary Outcome: Self-reported Functional Scores
Description: The percentage score of the Foot and Ankle Ability Measure (FAAM). The total percentage score ranges from 0-100. The higher score indicates a better ankle function.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percentage of FAAM
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 9 | 6
Percentage of FAAM | 82.8 (15.2) | 89.5 (13.8)

6. Secondary Outcome: Self-reported Functional Scores
Description: as for outcome 5
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Percentage of FAAM
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 9 | 6
Percentage of FAAM | 90.3 (15.4) | 98.4 (1.2)

7. Secondary Outcome: Spinal Reflex Excitability
Description: The maximal peak-to-peak amplitude ratios of the Hoffman reflex (H-reflex) and the motor response (M-wave) of the soleus muscle were calculated by normalizing the maximal H-reflex amplitude to the maximal M-wave amplitude (Hmax/Mmax ratio). A higher Hmax/Mmax indicates a greater spinal reflex excitability.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 8 | 5
Ratio | 0.40 (0.21) | 0.39 (0.10)

8. Secondary Outcome: Spinal Reflex Excitability
Description: as for outcome 7
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 8 | 5
Ratio | 0.40 (0.16) | 0.40 (0.18)

9. Secondary Outcome: Corticospinal Excitability as Evaluated by the Peak-to-peak Amplitude of Motor Evoked Potential (MEP)
Description: The soleus active muscle response, due to transcranial magnetic stimulation (TMS) pulses over the motor cortex, will be used for quantifying the motor evoked potential.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 8 | 5
mV | 0.68 (0.33) | 0.63 (0.25)

10. Secondary Outcome: Corticospinal Excitability as Evaluated by the Peak-to-peak Amplitude of Motor Evoked Potential (MEP)
Description: as for outcome 9
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 8 | 5
mV | 0.46 (0.16) | 0.46 (017)

11. Secondary Outcome: Dynamic Postural Control as Measured by the Reach Distance
Description: The anterior reach distance (cm) was measured by the Star Excursion Balance Test (SEBT).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 9 | 6
cm | 57.0 (3.6) | 55.9 (3.7)

12. Secondary Outcome: Dynamic Postural Control as Measured by the Reach Distance
Description: The anterior reach distance (cm) was measured by the Star Excursion Balance Test (SEBT).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 9 | 6
cm | 61.7 (4.5) | 62.2 (9.1)

13. Secondary Outcome: Dynamic Postural Balance as Measured by the Time to Complete the Lateral Hop
Description: The completion time (seconds) for the lateral hop will be measured. Each trial consists of 10 lateral hops. The average completion time of 3 trials will be reported. The completion time will be recorded using a stopwatch in seconds.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 9 | 6
second | 7.4 (2.9) | 7.2 (2.7)

14. Secondary Outcome: Dynamic Postural Balance as Measured by the Time to Complete the Lateral Hop
Description: as for outcome 13
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
Number analyzed (Participants) | 9 | 5
second | 5.3 (1.3) | 6.7 (3.8)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Anodal tDCS and Balance Training (BT) Group | Sham tDCS and BT Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT04390048/Prot_SAP_000.pdf